CLINICAL TRIAL: NCT03317691
Title: Automatic Diagnosis of ST-segment Elevated Myocardial Infarction by Artificial Intelligence-based Electrocardiographic System:The ALERT-Pilot Study
Brief Title: The ALERT-Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Professor, Shanghai 10th People's Hospital
Other Study IDs: 2017YFC0111800
Record Dates: First submitted 2017-10-12; First posted 2017-10-23 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Myocardial Infarction, Acute; Artificial Intelligence; ECG Pattern
Keywords: myocardial infarction; artificial Intelligence; 12 lead electrocardiogram
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ST segment Elevation Myocardial Infarction: ST segment Elevation Myocardial Infarction patients' diagnosis was confirmed by coronary artery angiography. The prior surgery electrocardiogram need to be collected.
  Interventions: Diagnostic Test: electrocardiogram diagnosed by artificial intelligence

INTERVENTIONS:
Diagnostic Test: electrocardiogram diagnosed by artificial intelligence — According to coronary angiogram results, the accuracy of STEMI patients' electrocardiogram diagnosis by artificial intelligence was evaluated.

SUMMARY:
the algorithm of artificial intelligent to diagnose myocardial infarction through prior surgery Electrocardiogram was established. The accuracy of using artificial intelligent to diagnose acute ST-segment elevation myocardial infarction and judge criminal vascular was evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. age≥18 years old;
2. the admitting doctor's diagnosis is ST-segment Elevation Myocardial Infarction.

Exclusion Criteria:

1. the admitting diagnosis is non-ST-segment Elevation Myocardial Infarction.
2. default data;
3. pregnancy, mental disorder, kidney failure;
4. except for criteria mention above, including some improper condition considered by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ST segment Elevation Myocardial Infarction patients' diagnosis was confired by coronary artery angiography. The prior surgery electrocardiogram need to be collected.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-10-15 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
the algorithm of artificial intelligent to diagnose myocardial infarction through prior surgery Electrocardiogram | 24 hours
  All the electrocardiograms done before coronary arteriography were read by artificial intelligent. Then according to results of coronary angiogram, artificial intelligent can establish a algorithm of to diagnose myocardial infarction.
The accuracy of using artificial intelligent to diagnose acute ST-segment elevation myocardial infarction and judge criminal vascular | 24 hours
  The accuracy of using artificial intelligent to diagnose acute ST-segment elevation myocardial infarction and judge criminal vascular was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided